CLINICAL TRIAL: NCT05791877
Title: Non-Invasive Measurement of Pulmonary Dysfunction in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Tariq Rahman, Principal Research Engineer, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1993376
Record Dates: First submitted 2023-03-09; First posted 2023-03-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Prospective observational study with a single group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cerebral palsy group (Experimental): Respiratory sensor will measure breathing in patients with Cerebral palsy
  Interventions: Device: pneuRIP

INTERVENTIONS:
Device: pneuRIP — Respiratory sensor to measure pulmonary function

SUMMARY:
This proposal addresses pulmonary dysfunction in severe cerebral palsy by using a novel non-invasive respiratory sensor. The two aims of the project are to 1) provide a screening tool to detect respiratory distress and 2) Find a correlation between the degree of pulmonary dysfunction and scoliosis in children with cerebral palsy.

DETAILED DESCRIPTION:
This project proposes the utilization of a novel non-invasive real-time breathing sensor - pneuRIP- to measure pulmonary function (PF) in children with high-level cerebral palsy. Currently the standard measures of PF such as spirometry and peak flow meters are too strenuous for children and those with severe CP, as a result they have low compliance rates. The pneuRIP does not require active user participation and can passively measure PF. It consists of two inductive bands worn around the chest and abdomen that measure and differentiate diaphragmatic and chest breathing through Respiratory Inductance Plethysmography (RIP). Readings are recorded and analyzed on a small chest-worn unit and wirelessly transmitted to an iPad. The pneuRIP yields indices of work of breathing (WOB) which includes the phase angle between the chest and abdomen; percentage breathing through the ribcage; respiratory rate; and labored breathing index. This sensor takes little time to set up and readings are provided instantaneously.

The WOB indices provide a screening tool for pulmonary diagnosis and treatment, decrease the risk for pneumonia and respiratory illness, and has the potential to act as a marker for scoliosis in children with high-level CP.

The impact on the field will be to have a simple and fast way to measure pulmonary function in children and adults with severe CP and correlate this to measures of function and scoliosis severity as the effects of scoliosis, which is common in CP, on pulmonary function is unclear. Measures of motor function are classified by the Gross Motor Functional Classification System (GMFCS), ranking from I to V, with worsening disability from near normal gait in Type I to complete wheelchair use in Type V. This project will address GMFCS levels IV and V which includes people using wheelchairs. The two specific aims are a) Measure WOB indices non-invasively using the pneuRIP sensor in children with CP who use a wheelchair (GMFCS level IV, V) and validate the use of WOB indices as a screening test for pulmonary dysfunction., 2) Determine the correlation between WOB indices and the degree of scoliosis using the pneuRIP sensor in 250 children with CP who use a wheelchair (GMFCS level IV, V).

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have cerebral palsy a GMFCS levels IV, V

Exclusion Criteria:

-

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Presence of pulmonary dysfunction | 1 month
  The presence of pulmonary dysfunction will be recorded for each subject. Presence will be determined clinically by the physician. Pulmonary dysfunction can take the form of pneumonia, ineffective airway clearance or atelectasis.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Rahman, PhD, Principal Investigator — Principal Research Engineer
Locations (1):
- Nemours Children's Hospital, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No